CLINICAL TRIAL: NCT06984471
Title: Characteristics of Patients in the ICU With Palliative Care Consults in a Tertiary University Hospital
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-00734; am25Sutter4
Record Dates: First submitted 2025-05-08; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Palliative Care Referral
Keywords: Intensive Care Unit

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Before ICU stay: Adult patients with a PC consult before an ICU stay at the University Hospital Basel between 2019 and until the end of 2024.
  Interventions: Other: Palliative care consult
- During ICU stay: Adult patients with a PC consult during an ICU stay at the University Hospital Basel between 2019 and until the end of 2024.
  Interventions: Other: Palliative care consult
- After ICU stay: Adult patients with a PC consult after an ICU stay at the University Hospital Basel between 2019 and until the end of 2024.
  Interventions: Other: Palliative care consult

INTERVENTIONS:
Other: Palliative care consult — A palliative care (PC) consult involves a specialized palliative care team to provide symptom management, psychosocial support, and assistance with goals-of-care discussions for patients with serious or life-limiting illnesses.

SUMMARY:
The aim of this retrospective observational single-center cohort study is to investigate the factors associated with palliative care (PC) referral, examine intensive care unit (ICU) involvement before, during, or after the referral, and evaluate patient outcomes such as mortality, hospital and ICU length of stay, discharge destination, functional status, symptom management, and the content of PC consultation reports.

DETAILED DESCRIPTION:
Palliative care (PC) in the intensive care unit (ICU) can improve care for critically ill patients by supporting decision-making, managing symptoms, and planning for end-of-life care. Early referral to PC has been linked to more do-not-resuscitate and do-not-intubate decisions, fewer ICU procedures, and more transfers to hospice care. However, PC is still underused in many ICUs, partly because doctors often overestimate patient survival. Most referral guidelines are based on older patients or those with serious conditions, which may not apply to younger or potentially recovering patients.

Existing studies mostly focus on survival or length of stay, with limited information on symptoms, functional recovery, or patient comfort. Some research suggests that PC needs are often not well met in the ICU.

This retrospective single-center cohort study aims to better understand when and why ICU patients are referred to PC, how their care changes, and what outcomes follow. It will also examine symptom management, functional outcomes, and recommendations made by the PC team.

The results of this study may help improve the timing and use of PC in the ICU to better support patient needs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (i.e., patients ≥18 years of age)
* Palliative care consult either before, during or after a ICU stay at the University Hospital Basel between 2019 and until the end of 2024

Exclusion Criteria:

* Patients younger than 18 years
* Patients with documented refusal to use data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive adult patients (i.e. >= 18 years of age) that received a palliative care consult in the same hospitalization as their ICU stay at the University Hospital Basel between 2019 and until the end of 2024. .
Sampling Method: Probability Sample
Enrollment: 532 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Patient demographics | 2019-2024
  Demographic information (e.g. age, sex) is collected.
Acute prehospital management data | 2019-2024
  Data from acute prehospital management, as documented in emergency medical services (EMS) treatment protocols, is collected. The collected data elements are aggregated to describe the overall EMS response.
Duration of intensive care unit stay | 2019-2024
  The length of intensive care unit (ICU) stay is recorded.
Duration of hospital stay | 2019-2024
  The length of the total hospital stay is recorded.
Discharge destination | 2019-2024
  The destination at discharge is recorded.
Date of palliative care consult | 2019-2024
  The specific date of palliative care consult is documented.
Reason for palliative care consult | 2019-2024
  The documented reason for palliative care consult is analyzed.
Place of palliative care consult | 2019-2024
  The specific place of palliative care consult is documented.
Number of visits by the palliative care team | 2019-2024
  The number of visits by the palliative care team is analyzed.
Additional features of the palliative care consult | 2019-2024
  Assessment of additional features related to the palliative care consult (changes in management, referral for psychiatric or psychological evaluation, treatment recommendations, etc.) documented in the medical records or consult report. These features are aggregated to characterize the scope, complexity, and potential impact of the palliative care consultation on the patient's overall treatment and care trajectory.
Comprehensive assessment of the neurological status based on validated clinical assessment | 2019-2024
  Neurological status during ICU stay is assessed using available data in the patient register from validated neurological assessments. These may include the Richmond Agitation-Sedation Scale (RASS), Sedation-Agitation Scale (SAS), Glasgow Coma Scale (GCS), Intensive Care Delirium Screening Checklist (ICDSC), or Status Epilepticus Severity Score (STESS). The specific tool used, as well as the scale of the score and meaning behind the score, depends on routine clinical practice and available documentation in the register. If multiple scores are available for a patient, they will be aggregated to provide a comprehensive assessment of neurological status. This outcome will be reported as a descriptive summary, synthesizing findings across tools, rather than as a single quantitative score.
Comprehensive assessment of critical illness severity based on standardized scoring systems | 2019-2024
  Disease severity during ICU stay is assessed using standardized scoring systems, including the Acute Physiology and Chronic Health Evaluation II (APACHE II), Simplified Acute Physiology Score II (SAPS II), and Sequential Organ Failure Assessment (SOFA), depending on data availability in the patient register. The specific scoring system applied, as well as the scale and interpretation of the score, varies based on routine clinical practice and available documentation. Where multiple severity scores are available, they will be synthesized to provide a descriptive summary of overall illness severity rather than a single quantitative score.
Charlson Comorbidity Index | 2019-2024
  The Charlson Comorbidity Index (CCI) is calculated based on pre-existing comorbidities and additional diagnoses. The CCI predicts the ten-year mortality for a patient who may have a range of comorbid conditions. It assigns weighted scores (from 0 to maximal 6) to 17 comorbid conditions (e.g., heart disease, diabetes, cancer), resulting in a total score ranging from 0 to 33, if the patient had the most severe form of each of the 17 conditions.
Laboratory parameters | 2019-2024
  Routine laboratory value for e.g. C-Reactive Protein (CRP), albumin, Lactate Dehydrogenase (LDH), Creatine Kinase (CK), procalcitonin, white blood cell levels, creatinine, liver enzymes, blood gas analyses, metabolic data, etc. is collected. The specific parameters recorded may vary depending on the laboratory assessments documented in the patient register. All values will be reported using their respective units of measurement.These parameters are aggregated to support an overall clinical interpretation rather than a single numerical value. This approach reflects standard clinical practice, where multiple lab values are considered together to assess a patient's condition.
Complications associated with palliative Care consult | 2019-2024
  The complications occurring during or after the palliative care consultation are recorded, including inadequate symptom control, dissatisfaction expressed by the patient or relatives, cardiac arrest, unplanned emergency transfers to the ICU, and poor functional outcomes.
Glasgow Outcome Score | 2019-2024
  The Glasgow Outcome Score (GOS) is calculated based on the assessment of key clinical outcomes such as inhospital mortality, survival, survival with neurofunctional alteration, return to premorbid neurological function, and hospital readmission to determine the patient outcome.
  The GOS ranges from 1 (death) to 5 (good recovery).
Therapeutic intervention | 2019-2024
  The therapeutic intervention is documented, including information on duration, dosage and number of treatment medication, number of neuroleptic, sedative and analgesic drugs, invasive procedures, such as intubation, mechanical, ventilation, vasopressors, installation of central lines, nutrition, etc.
Vital signs | 2019-2024
  Vital signs are analyzed based on the data available in the patient register. These may include blood pressure, heart rate, respiratory rate, oxygen saturation, body temperature, level of consciousness, etc. The specific parameters recorded depend on the clinical documentation available. All values will be reported using their respective units of measurement. These values are aggregated to support an overall clinical assessment rather than a single numerical score. This reflects standard practice, where multiple vital signs are interpreted together to evaluate a patient's condition.
Fluid balance data | 2019-2024
  Fluid balance data, including the administration of fluids such as blood products, crystalloids, and enteral/parenteral nutrition, are documented. These components are aggregated to represent overall fluid input for each patient.
Assessment of diagnostic procedure | 2019-2024
  The diagnostic procedures performed during intensive care-whether invasive (e.g., lumbar puncture, central line placement) or non-invasive (e.g., radiologic imaging, ultrasound)-are systematically documented. Additionally, if physical restraints are used to ensure patient safety or procedural success, their usage are also recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Raoul Sutter, Prof. Dr. med., Principal Investigator — University Hospital Basel, Clinic for Intensive Care Medicine
Locations (1):
- University Hospital Basel, Clinic for Intensive Care Medicine, Basel, Switzerland